CLINICAL TRIAL: NCT00590876
Title: The Impact of Pancreatic Islet Cell Allotransplantation on Cognitive Function and Brain Fuel Utilization in Patients With Type 1 Diabetes and Hypoglycemia Unawareness
Brief Title: The Impact of Pancreatic Islet Cell Allotransplantation on Cognitive Function in Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Robert Sherwin, CNH Long Professor, Yale University
Other Study IDs: DK66108a_0304025134; R37DK020495 (NIH); DK20495
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Hypoglycemia; Pancreatic Islet Cell Allotransplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: T1DM patients with a history of severe hypoglycemia and/or hypoglycemia unawareness who have been selected based upon this history to undergo islet cell transplantation at the University of Minnesota.
- 2: T1DM patients (C-peptide negative) who are matched for age, gender, and duration of diabetes, who also have a history of severe hypoglycemia and/or hypoglycemia unawareness meeting the criteria for islet cell transplantation. The hemoglobin A1c for each of these subjects will fall within 1% of the islet transplant recipient to whom they are matched.
- 3: Nondiabetic subjects (fasting plasma glucose < 110 mg/dl) who are matched for age and gender to the islet transplant recipient to whom they are matched.

SUMMARY:
In patients with Type 1 Diabetes Mellitus, hypoglycemia (low blood sugar) is the rate-limiting step to achieve glucose level control. As a result, understanding the body's responses (including the brain's response) to hypoglycemia is essential for the effective treatment of patients with T1DM. The purpose of this research is to determine whether pancreatic islet cell allotransplantation to restore normoglycemia (normal blood glucose levels) in Type 1 Diabetic patients with hypoglycemia unawareness alters brain fuel utilization and cognitive performance under euglycemic (blood sugar at 100 mg/dl) and hypoglycemic (blood sugar at 50 mg/dl) conditions. Three groups of subjects will be studied: (1) T1DM patients with a history of severe hypoglycemia and/or hypoglycemia unawareness who have been selected for pancreatic islet cell allotransplantation; (2) T1DM patients who also have a history of severe hypoglycemia and/or hypoglycemia unawareness; (3) nondiabetic subjects. All subjects will undergo identical testing including: (a) screening; (b) neuropsychological testing; (c) and functional magnetic resonance imaging (fMRI) during euglycemic and hypoglycemic conditions.

ELIGIBILITY:
Inclusion Criteria:

* T1DM subjects must be 18 years or older and able to provide written consent
* T1DM subjects must be undergoing intensive management, defined by self-monitoring of glucose values 3 or more times each day and by the administration of 3 or more insulin injections each day (or the use of insulin pump therapy). This clinical management must be monitored in close cooperation with an endocrinologist as defined by at least 3 contacts during the previous 12 months.
* T1DM subjects must demonstrate at least one of the following situations that persist despite intensive insulin management efforts:
* metabolic lability/instability, characterized by either 2 or more episodes of severe hypoglycemia within one year (defined as an event with symptoms consistent with hypoglycemia in which the patient requires the assistance of another person, and which is associated with a blood glucose of < 50 mg/dl or prompt recovery after administration of oral carbohydrate, intravenous glucose, or glucagon) or 2 or more hospital admissions for diabetic ketoacidosis over the last year.
* reduced awareness of hypoglycemia (defined by a specific hypoglycemia questionnaire)

Exclusion Criteria:

* Age < 18 years
* Body weight > 75 kg at screening
* BMI > 24 (female) and > 25 (male) kg/m2
* Waist to hip ratio greater than or equal to 0.80 (female) and greater than or equal to 0.95 (male)
* Insulin requirement of > 0.7IU/kg/day or > 50 IU per day, whichever is less
* Positive C-peptide response to intravenous arginine stimulation (5g): any C-peptide greater than or equal to 0.2ng/ml at 2, 3, 4, 5, 7, and 10 minutes post infusion
* Untreated proliferative retinopathy
* Creatinine clearance < 75ml/min/1.73 m2
* Serum creatinine greater than or equal to 1.3 mg/dl for females, and greater than or equal to 1.5 mg/dl for males
* Previous pancreas or islet cell transplant
* Presence of history of panel-reactive anti-HLA antibodies > 10%
* Positive pregnancy test or presently breast-feeding, or failure to follow effective contraceptive measures or abstinence (oral contraceptives, Norplant, Depo-Provera, and barrier devices are acceptable; condom use alone is not acceptable.)
* Active infection including Hepatitis C, Hepatitis B, HIV, or Tuberculosis (or under treatment for suspected Tuberculosis)
* Negative screen for Epstein-Barr Virus (EBV) or by an EBNA method
* Invasive aspergillus infection within a year prior to study entry
* Any history of malignancy except for adequately treated squamous cell or basal cell carcinoma of the skin
* Active alcohol or substance abuse which includes cigarette smoking (must be abstinent for 6 months). Active alcohol use abuse should be considered using the current NIAAA definitions whereby alcohol abuse is defined by a pattern of drinking that is accompanied by one or more of the following situations within a 12-month period:
* Failure to fulfill major work, school, or home responsibilities
* Drinking in situations that are physically dangerous, such as while driving a car or operating machinery
* Recurring alcohol-related legal problem, such as being arrested for driving under the influence of alcohol or for physically hurting someone while drunk
* Continued drinking despite having ongoing relationship problems that are caused or worsened by the effects of alcohol
* History of nonadherence to prescribed regimens
* Psychiatric disorder making the subject not a suitable candidate for transplantation (for those who are undergoing islet cell allotransplantation).
* Inability to provide informed consent
* Baseline Hgb < 11.7 g/dl in females, or < 13 g/dl in males; lymphopenia (< 1 ,000 lymphocytes/mcl) or leukopenia (< 3,000 total leukocytes/mcl), or an absolute CD4 count < 500, or platelets < 150,000
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g. warfarin) after transplantation (low-dose aspirin treatment is allowed) or patient with INR > 1.5
* Severe co-existing cardiac disease, characterized by any one of the following conditions:
* recent myocardial infarction (within the past 6 months) or
* angiographic evidence of non-correctable coronary artery disease, or
* evidence of ischemia on functional cardiac exam (to be repeated annually)or
* left ventricular ejection fraction < 30%
* Baseline liver function tests outside of normal range or a history of significant liver disease
* Presence of gallstones or hemangioma in the liver on baseline ultrasound exam
* Active peptic ulcer disease
* Severe unremitting diarrhea or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
* Presence of severe allergy requiring acute (within 4 weeks of baseline), or chronic treatment
* Known hypersensitivity to rabbit proteins
* Hyperlipidemia (fasting LDL cholesterol > 139 mg/dl, treated, or untreated; and/or fasting triglycerides > 200 mg/dl
* Addison's Disease
* Under treatment for a medical condition requiring chronic use of systemic steroids
* Any medical condition that, in the opinion of the investigators, will interfere with the safe completion of the study
* Presence of implanted ferromagnetic devices

Inclusion criteria for nondiabetic control subjects:

* Fasting glucose < 110 mg/dl and otherwise healthy
* Age > 18 years
* Body weight parameters the same as for subjects with diabetes (above)

Exclusion criteria for nondiabetic control subjects:

* Pregnancy or presently breastfeeding or failure to follow effective contraceptive measures including abstinence (as noted above)
* Active alcohol or substance abuse (as defined above)including cigarettes. Must be abstinent of tobacco for 6 months
* Psychiatric disorder making the subject not suitable for following the protocol
* Presence of implanted ferromagnetic devices

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing pancreatic islet cell allotransplantation at the University of Minnesota
  Patients who are seen at Diabetes Clinics at Yale School of Medicine
  Nondiabetic, healthy subjects from New Haven and surrounding communities
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
fMRI | 0, 3, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Minnesota, Minneapolis, Minnesota